CLINICAL TRIAL: NCT06811740
Title: The Study About the Identification of Treatable Traits of Severe Asthma and the Construction of Personalized Treatment System
Brief Title: Treatable Traits of Severe Asthma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Capital Medical University (Other); Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Kewu Huang, Professor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KE-338
Record Dates: First submitted 2025-02-05; First posted 2025-02-06 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: treatable traits; asthma; severe; AQLQ; ACQ
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Implement individualized cluster management based on treatable traits
  Interventions: Procedure: Individualized cluster management
- Placebo (Other): Routine asthma treatment according to current guidelines
  Interventions: Procedure: Routine asthma treatment

INTERVENTIONS:
Procedure: Individualized cluster management — Individualized cluster management for treatable traits
  Arms: Intervention group
Procedure: Routine asthma treatment — Routine asthma treatment according to current guidelines
  Arms: Placebo

SUMMARY:
Severe or uncontrolled asthma is a complex heterogeneous disease, in which patients may exhibit different types of airway inflammation and often accompany multiple comorbidities and risk factors. Identifying potential modifiable factors that influence prognosis, i.e., "treatable traits," and targeting these traits for individualized, bundled management of patients may help improve the quality of life of asthma patients and enhance asthma control levels. This project aims to investigate the distribution of treatable traits in uncontrolled asthma patients in Beijing by conducting pulmonary function tests, exhaled nitric oxide tests, blood tests, allergen IgE tests, and chest CT scans, as well as detailed questionnaires, on patients from three tertiary hospitals in Beijing. The project will also assess the impact of treatable traits on the quality of life or asthma control levels of uncontrolled asthma patients in a multidimensional manner. Furthermore, the project will select severe asthma patients and establish an individualized, bundled management model based on the treatable traits of severe asthma, through multidisciplinary consultations and shared decision-making with patients. A randomized, parallel-group clinical trial will then be conducted for six months to confirm whether this management model is superior to conventional management in improving the quality of life or asthma control levels of severe asthma patients. The implementation of this project will establish a new model of individualized management for severe asthma based on treatable traits, thereby improving the management level of severe asthma.

ELIGIBILITY:
Inclusion Criteria

* Must be at least 18 years old and have resided in Beijing for at least 6 months.
* Must meet the diagnostic criteria for asthma as outlined in the 2023 GINA guidelines, have written evidence of variable airflow limitation, and have been receiving asthma treatment for at least 6 months.
* Must meet one or both of the following criteria as defined in the 2023 GINA guidelines for uncontrolled asthma: poor symptom control (defined as an Asthma Control Questionnaire (ACQ-5) score of 0.75 or higher); frequent acute exacerbations (≥2 per year) requiring oral corticosteroids, or severe acute exacerbations (≥1 per year) requiring emergency or hospitalization.
* Willing to undergo a multidisciplinary, multi-dimensional evaluation and sign an informed consent form.
* Must meet the criteria for severe asthma as outlined in the 2023 GINA guidelines

Exclusion Criteria

* Use macrolides within 4 weeks of the screening period
* Use anti-IgE, anti-IL-5, or anti-IL-5R therapy within 4 weeks of the screening period
* Use inhaled ICS + LABA + long-acting muscarinic antagonist (LAMA) within 4 weeks of the screening period
* Be allergic to macrolides
* Have a QTc interval prolongation of >480ms
* Take a medication that interacts with azithromycin to prolong the QTc interval or cause existing ECG abnormalities, which may lead to arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Quality of life score (AQLQ) | 6 months
  Changes in asthma Quality of life score (AQLQ) from baseline at 6 months；Asthma Quality of Life questionnaire (AQLQ) is a scoring scale to evaluate the quality of life of patients with asthma, evaluating the level of asthma control in the past 2 weeks. The AQLQ consisted of 32 questions, which were divided into four sub-areas: symptoms (12 questions), activity limitation (11 questions), emotional function (5 questions) and environmental stimulation (4 questions). Each question was scored on a scale of 1 to 7 points according to its severity, with 1 indicating complete limitation and 7 indicating no limitation at all. The total score is calculated as the average of all questions and the average of each partition.

SECONDARY OUTCOMES:
Asthma Control Questionnaire score (ACQ-5) | 6 months
  Changes in Asthma Control Questionnaire score (ACQ-5) from baseline at 6 months；ACQ-5 (Asthma Control Questionnaire) is a scoring scale for assessing asthma control. It consists of 5 simple questions to assess a patient's level of asthma control in the past week. Each problem was scored on a scale of 0-6 according to its severity. The average score of the five problems <0.75 was asthma control, 0.75 ~ 1.5 was asthma partial control, and >1.5 was asthma uncontrolled.
Forced Expiratory Volume in 1 second（FEV1） | 6 months
  Changes in lung function Forced Expiratory Volume in 1 second（FEV1） from baseline
Exacerbation | 6 months
  the number of acute asthma attacks within 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Institute of Respiratory Medicine and Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Haidian
  - Beijing Luhe Hospital affiliated to Capital Medical University, Beijing, Tongzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rose L, Istanboulian L, Carriere L, Thomas A, Lee HB, Rezaie S, Shafai R, Fraser I. Program of Integrated Care for Patients with Chronic Obstructive Pulmonary Disease and Multiple Comorbidities (PIC COPD+): a randomised controlled trial. Eur Respir J. 2018 Jan 11;51(1):1701567. doi: 10.1183/13993003.01567-2017. Print 2018 Jan. PMID 29326330
- [Background] Ko FW, Cheung NK, Rainer TH, Lum C, Wong I, Hui DS. Comprehensive care programme for patients with chronic obstructive pulmonary disease: a randomised controlled trial. Thorax. 2017 Feb;72(2):122-128. doi: 10.1136/thoraxjnl-2016-208396. Epub 2016 Jul 28. PMID 27471050
- [Background] McDonald VM, Fingleton J, Agusti A, Hiles SA, Clark VL, Holland AE, Marks GB, Bardin PP, Beasley R, Pavord ID, Wark PAB, Gibson PG; participants of the Treatable Traits Down Under International Workshop; Treatable Traits Down Under International Workshop participants:. Treatable traits: a new paradigm for 21st century management of chronic airway diseases: Treatable Traits Down Under International Workshop report. Eur Respir J. 2019 May 9;53(5):1802058. doi: 10.1183/13993003.02058-2018. Print 2019 May. PMID 30846468
- [Background] Wu WW, Zhang X, Li M, Liu Y, Chen ZH, Xie M, Zhao SZ, Wang G, Zhang HP, Wang T, Qin L, Wang L, Oliver BG, Wan HJ, Zhang J, McDonald VM, Marks GB, Li WM, Birring SS, Wang G, Gibson PG. Treatable Traits in Elderly Asthmatics from the Australasian Severe Asthma Network: A Prospective Cohort Study. J Allergy Clin Immunol Pract. 2021 Jul;9(7):2770-2782. doi: 10.1016/j.jaip.2021.03.042. Epub 2021 Apr 5. PMID 33831621
- [Background] McDonald VM, Hiles SA, Godbout K, Harvey ES, Marks GB, Hew M, Peters M, Bardin PG, Reynolds PN, Upham JW, Baraket M, Bhikoo Z, Bowden J, Brockway B, Chung LP, Cochrane B, Foxley G, Garrett J, Jayaram L, Jenkins C, Katelaris C, Katsoulotos G, Koh MS, Kritikos V, Lambert M, Langton D, Lara Rivero A, Middleton PG, Nanguzgambo A, Radhakrishna N, Reddel H, Rimmer J, Southcott AM, Sutherland M, Thien F, Wark PAB, Yang IA, Yap E, Gibson PG. Treatable traits can be identified in a severe asthma registry and predict future exacerbations. Respirology. 2019 Jan;24(1):37-47. doi: 10.1111/resp.13389. Epub 2018 Sep 19. PMID 30230137
- [Background] McDonald VM, Clark VL, Cordova-Rivera L, Wark PAB, Baines KJ, Gibson PG. Targeting treatable traits in severe asthma: a randomised controlled trial. Eur Respir J. 2020 Mar 5;55(3):1901509. doi: 10.1183/13993003.01509-2019. Print 2020 Mar. PMID 31806719
- See also: Related Info — https://ginasthma.org/2023-gina-main-report/